CLINICAL TRIAL: NCT01686646
Title: Effects of Two Doses of a Common Cold Treatment on Cognitive Function
Brief Title: Effects of Two Doses of a Common Cold Treatment on Alertness
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RH01361
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Results first posted 2014-07-14 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-07

CONDITIONS: Common Cold
Keywords: alertness
MeSH Terms: conditions — Common Cold | interventions — Acetaminophen; Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- highest dose Paracetamol + caffeine (Active Comparator): highest dose of Paracetamol and caffeine
  Interventions: Drug: paracetamol + caffeine
- low-dose Paracetamol + caffeine (Active Comparator): lowest dose of Paracetamol and caffeine
  Interventions: Drug: paracetamol + caffeine
- high dose paracetamol (Active Comparator): highest dose paracetamol
  Interventions: Drug: paracetamol
- low dose paracetamol (Active Comparator): lowest dose paracetamol
  Interventions: Drug: paracetamol

INTERVENTIONS:
Drug: paracetamol + caffeine — paracetamol with caffeine
  Arms: highest dose Paracetamol + caffeine; low-dose Paracetamol + caffeine
Drug: paracetamol — paracetamol
  Arms: high dose paracetamol; low dose paracetamol

SUMMARY:
This study will investigate any improvement in alertness and performance based on cognitive function and mood assessment in subjects suffering the common cold, when taking a novel paracetamol and caffeine combination verses paracetamol alone.

ELIGIBILITY:
* Participants with symptoms of cold < 96 hours, rating of at least '2' on malaise at least 4 other symptoms of cold.
* No history of clinically significant perennial rhinitis, no recent antibiotic, antihistamine or cold treatment, no caffeine in the previous 12 hours, no psychoactive medication in the 14 days prior to screening, no pregnancy, breastfeeding or participation in this trial, or another trial in the 30 days prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Common Cold Centre, Cardiff, Wales, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site.
Pre-assignment Details: Out of 244 participants screened, 4 did not meet the study criteria. Remaining 240 were randomized into the study.
Groups:
- Paracetamol + Caffeine Combination (1000/130): Two paracetamol (500 milligrams [mg] ) and caffeine (65 mg) tablets were dissolved in 200 milliliter (mL) of water and administered orally.
- Paracetamol (1000): Two paracetamol tablets (500 mg each) were dissolved in 200 mL of water and administered orally.
- Paracetamol + Caffeine Combination (500/65): One paracetamol (500 mg) and caffeine (65 mg) tablet was dissolved in 200 mL of water and administered orally.
- Paracetamol (500): One paracetamol tablet (500 mg) was dissolved in 200 mL of water and administered orally.
Period: Overall Study
Arm/Group | Paracetamol + Caffeine Combination (1000/130) | Paracetamol (1000) | Paracetamol + Caffeine Combination (500/65) | Paracetamol (500)
Started | 45 | 45 | 75 | 75
Intent to Treat Population | 45 | 45 | 75 | 75
Safety Population | 46 (One subject randomized to Paracetamol+Caffeine (500/65) group but received 1000/130 combination.) | 45 | 74 | 75
Completed | 45 | 45 | 75 | 75
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Paracetamol + Caffeine Combination (1000/130): Two paracetamol (500 mg) and caffeine (65 mg) tablets were dissolved in 200 mL of water and administered orally.
- Total: Total of all reporting groups
Arm/Group | Paracetamol + Caffeine Combination (1000/130) | Paracetamol (1000) | Paracetamol + Caffeine Combination (500/65) | Paracetamol (500) | Total
Number analyzed (Participants) | 46 | 45 | 74 | 75 | 240
Age, Continuous [Mean (Standard Deviation); unit: Years] | 20.0 (1.56) | 20.0 (1.74) | 20.6 (4.19) | 20.2 (2.80) | 20.2 (2.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 28 | 47 | 48 | 154
  Male | 15 | 17 | 27 | 27 | 86

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Number of Accurate Responses to Rapid Visual Information Processing (RVIP) Cognitive Test
Description: The RVIP assessed the performance of visual attention mechanisms in remaining vigilant to periodically occurring events. The number of accurate responses to RVIP task was determined from the cognitive function computerised output. Participants monitored a series of single numbers (0-9) appearing in the centre of the screen. During the RVIP task, participants responded to consecutive sequences of three odd or three even numbers by pressing the corresponding response button as quickly and accurately as possible. This was identified in the output file by a value of '1' in 'TARGET=1' column. Also, the response time (in seconds) was recorded in the 'RT' column. If the subject correctly responded to the target, this was identified by a value of '1' in the 'CORRECT=1' column. The number of accurate responses was calculated as the total number of records where 'CORRECT=1' had a value of '1'. The test lasted approximately 9 minutes and number of accurate responses to stimulus was calculated.
Time Frame: Baseline to 60 minutes post treatment administration
Population: Intent to Treat (ITT) population: all randomized participants who received study treatment and had at least one post-baseline efficacy evaluation.
Measure: Least Squares Mean (Standard Error); unit: Correct responses
Arm/Group | Paracetamol + Caffeine Combination (1000/130) | Paracetamol (1000) | Paracetamol + Caffeine Combination (500/65) | Paracetamol (500)
Number analyzed (Participants) | 45 | 45 | 75 | 75
Correct responses | 8.3 (1.12) | 4.8 (1.12) | 4.5 (0.89) | 2.7 (0.88)
Statistical Analysis 1: Comparison: Paracetamol + Caffeine Combination (1000/130) vs Paracetamol (1000); Null hypothesis was no difference in treatments in the change from baseline in the number of valid responses from the RVIP; Test type: Superiority or Other; p = 0.0248, ANCOVA — A hierarchical testing procedure was used such that p-values were only presented if the preceding treatment comparison was statistically significant (p<0.05); From ANCOVA model with factors for treatment group and season, and baseline score as a covariate; LS Mean DIfference = 3.5, 95% CI 2-sided [0.4 to 6.5] — A positive difference favored the first named treatment
Statistical Analysis 2: Comparison: Paracetamol + Caffeine Combination (500/65) vs Paracetamol (500); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1513, ANCOVA — [p-value comment as in outcome 1, analysis 1]; From ANCOVA model with factors for treatment group and season, and baseline score as a covariate; LS Mean Difference = 1.7, 95% CI 2-sided [-0.6 to 4.1] — A positive difference favoured the first named treatment
Statistical Analysis 3: Comparison: Paracetamol + Caffeine Combination (1000/130) vs Paracetamol + Caffeine Combination (500/65); Null hypothesis was no difference in treatments in change from baseline in number of valid responses from RVIP task; Test type: Superiority or Other; ANCOVA — Not significant based on hierarchical testing; From ANCOVA model with factors for treatment group and season, and baseline score as a covariate; LS Mean Difference = 3.9, 95% CI 2-sided [1.1 to 6.6] — A positive difference favoured the first named treatment

2. Secondary Outcome: Change From Baseline in Number of Accurate Responses to RVIP Cognitive Test
Description: as for outcome 1
Time Frame: Baseline to 120 minutes post treatment administration
Population: ITT population: all randomized participants who received study treatment and had at least one post-baseline efficacy evaluation.
Measure: Least Squares Mean (Standard Error); unit: Correct responses
Arm/Group | Paracetamol + Caffeine Combination (1000/130) | Paracetamol (1000) | Paracetamol + Caffeine Combination (500/65) | Paracetamol (500)
Number analyzed (Participants) | 45 | 45 | 75 | 75
Correct responses | 7.3 (1.16) | 4.4 (1.15) | 6.2 (0.91) | 3.5 (0.92)
Statistical Analysis 1: Comparison: Paracetamol + Caffeine Combination (1000/130) vs Paracetamol (1000); Null hypothesis was no difference in treatments in the change from baseline in the number of accurate responses from the RVIP; Test type: Superiority or Other; p = 0.0696, ANCOVA — [p-value comment as in outcome 1, analysis 1]; From ANCOVA model with factors for treatment group and season, and baseline score as a covariate; LS Mean Difference = 2.9, 95% CI 2-sided [-0.2 to 6.1] — A positive difference favored the first named treatment
Statistical Analysis 2: Comparison: Paracetamol + Caffeine Combination (500/65) vs Paracetamol (500); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 1, analysis 1]; From ANCOVA model with factors for treatment group and season, and baseline score as a covariate; LS Mean Difference = 2.7, 95% CI 2-sided [0.3 to 5.2] — A positive difference favored the first named treatment
Statistical Analysis 3: Comparison: Paracetamol + Caffeine Combination (1000/130) vs Paracetamol + Caffeine Combination (500/65); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 1, analysis 1]; From ANCOVA model with factors for treatment group and season, and baseline score as a covariate; LS Mean Difference = 1.1, 95% CI 2-sided [-1.7 to 3.9] — A positive difference favored the first named treatment

3. Secondary Outcome: Change From Baseline in Mean Time of Accurate Responses to RVIP Cognitive Task
Description: The mean time of accurate responses was defined as the mean reaction time for the correct responses. For records with '1' in the 'CORRECT=1' column, the mean time of accurate response was calculated as the summation of the response time values divided by number of records with '1' in the 'CORRECT=1' column. The result was multiplied by 1000 to convert into milliseconds (msecs).
Time Frame: Baseline, 60 minutes and upto 120 minutes post treatment administration
Population: as for outcome 2
Measure: Median (Full Range); unit: milliseconds (msec)
Arm/Group | Paracetamol + Caffeine Combination (1000/130) | Paracetamol (1000) | Paracetamol + Caffeine Combination (500/65) | Paracetamol (500)
Number analyzed (Participants) | 45 | 45 | 75 | 75
milliseconds (msec)
  60 minutes | -1.4 [-92 to 102] | 2.4 [-113 to 313] | -0.9 [-134 to 119] | -9.9 [-108 to 142]
  120 minutes | -10.3 [-62 to 125] | -6.0 [-86 to 71] | -12.5 [-91 to 109] | -14.0 [-144 to 136]

4. Secondary Outcome: Change From Baseline in Number of Inaccurate and Missed Responses to RVIP Cognitive Task
Description: The no. of inaccurate responses to RVIP was determined from cognitive function computerised output. Participants monitored a series of single numbers (0-9) appearing in the centre of screen. They responded to consecutive sequences of 3 odd or even numbers by pressing the corresponding response button. This was identified in the output file by a value of '1' in the 'TARGET=1' column. If a subject responded incorrectly to stimuli (pressed the response button at the wrong time), this was identified by a value of '-1' in the 'CORRECT=1' column. The no. of incorrect responses was calculated as the total no. of records where 'CORRECT=1' had a value of '-1'. If the subject missed a target (failed to press the response button within 600 msecs of being presented with a string of 3 consecutive even or odd numbers), this was considered a missed response and was calculated as the no. of records where there was a value of '1' in the 'TARGET=1' column and a value of '0' in the 'CORRECT=1' column.
Time Frame: Baseline, 60 minutes and up to 120 minutes post treatment administration
Population: as for outcome 2
Measure: Mean (Standard Error); unit: inaccurate and missed responses
Arm/Group | Paracetamol + Caffeine Combination (1000/130) | Paracetamol (1000) | Paracetamol + Caffeine Combination (500/65) | Paracetamol (500)
Number analyzed (Participants) | 45 | 45 | 75 | 75
inaccurate and missed responses
  Incorrect responses at 60 minutes | -5.7 (3.43) | -2.8 (1.38) | 1.4 (1.96) | -2.4 (1.82)
  Incorrect responses at 120 minutes | -4.5 (4.12) | -1.7 (1.78) | -0.8 (1.97) | -3.3 (1.56)
  Missed responses at 60 minutes | -8.1 (1.03) | -4.8 (1.18) | -4.8 (0.83) | -3.1 (0.89)
  Missed responses at 120 minutes | -7.6 (1.14) | -4.8 (1.15) | -6.5 (0.80) | -3.5 (0.92)

5. Secondary Outcome: Change From Baseline in Number of Accurate Responses to Sustained Attention Tasks (SAT) Cognitive Test
Description: Auditory and visual attention of participants was evaluated using a validated Sustained Attention task. For the sustained auditory attention task, participants were required to respond whenever they heard the number '8' in a continuous stream of numbers presented through headphones. This was identified in the output file by a value of '8' in the 'NUMBER' column. For the sustained visual attention task, participants were required to respond to the letter 's' every time it appeared in a continuous stream of letters presented on a screen. This was identified in the output file by a value of 's' in the 'LETTER' column. If the subject correctly responded to the target, this was identified by a value of '1' in the 'CORRECT=1' column. The number of accurate responses was calculated as the total number of records where 'CORRECT=1' had a value of '1'.
Time Frame: Baseline, 60 minutes and up to 120 minutes post treatment administration
Population: as for outcome 2
Measure: Median (Full Range); unit: Correct responses
Arm/Group | Paracetamol + Caffeine Combination (1000/130) | Paracetamol (1000) | Paracetamol + Caffeine Combination (500/65) | Paracetamol (500)
Number analyzed (Participants) | 45 | 45 | 75 | 75
Correct responses
  Number of Accurate Responses to SAT at 60 mins | 1.0 [-4 to 16] | 0.5 [-16 to 43] | 2.0 [-9 to 33] | 0.0 [-28 to 15]
  Number of Accurate Responses to SAT at 120 mins | 2.0 [-17 to 28] | 1.0 [-11 to 42] | 1.0 [-6 to 30] | 2.0 [-10 to 26]

6. Secondary Outcome: Change From Baseline in Mean Time of Accurate Responses to SAT Cognitive Task
Description: as for outcome 3
Time Frame: Baseline, 30 minutes and up to 60 minutes post treatment administration
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | Paracetamol + Caffeine Combination (1000/130) | Paracetamol (1000) | Paracetamol + Caffeine Combination (500/65) | Paracetamol (500)
Number analyzed (Participants) | 45 | 45 | 75 | 75
msec
  60 minutes | -16.7 (3.17) | -9.8 (3.17) | -10.8 (2.51) | -12.0 (2.47)
  120 minutes | -21.2 (3.48) | -10.4 (3.48) | -18.0 (2.74) | -15.4 (2.72)

7. Secondary Outcome: Change From Baseline in Number of Incorrect and Missed Responses to SAT Cognitive Test
Description: For sustained auditory attention task, participants were required to respond on hearing the no. '8' in a continuous stream of numbers through headphones. It was identified in output file by a value of '8' in 'NUMBER' column. For sustained visual attention task, participants responded to letter 's' every time it appeared in a continuous stream of letters presented on screen. This was identified in output file by a value of 's' in 'LETTER' column. If a subject responded incorrectly (pressed the response button at the wrong time), it was identified by a value of '-1' in 'CORRECT=1' column. The no. of incorrect responses was calculated as total no. of records where 'CORRECT=1' had a value of '-1'. The no. of missed responses (when subject failed to press the response button on hearing the number '8' or seeing the letter 's'), was calculated as the no. of records where there was a value of '8' in 'NUMBER' column or 's' in the 'LETTER' column and a value of '0' in the 'CORRECT=1' column.
Time Frame: Baseline, 60 minutes and up to 120 minutes post treatment administration
Population: as for outcome 2
Measure: Mean (Standard Error); unit: incorrect and missed responses
Arm/Group | Paracetamol + Caffeine Combination (1000/130) | Paracetamol (1000) | Paracetamol + Caffeine Combination (500/65) | Paracetamol (500)
Number analyzed (Participants) | 45 | 45 | 75 | 75
incorrect and missed responses
  Incorrect responses at 60 minutes | -4.6 (1.00) | -1.1 (0.87) | -4.2 (0.74) | -1.6 (0.71)
  Incorrect responses at 120 minutes | -4.4 (1.04) | -2.3 (0.98) | -4.3 (0.88) | -2.8 (0.82)
  Missed responses at 60 minutes | -2.7 (0.74) | -1.9 (1.25) | -2.3 (0.70) | -0.8 (0.66)
  Missed responses at 120 minutes | -2.8 (1.11) | -2.0 (1.19) | -2.2 (0.64) | -2.4 (0.63)

8. Secondary Outcome: Change From Baseline in Number of Valid Responses to Divided Attention Task (DAT) Cognitive Test
Description: Auditory and visual attention of participants was evaluated using a validated Divided Attention task. Participants were required to respond whenever they heard the number '8' in a continuous stream of numbers presented through headphones or saw a letter 's' on the screen . This was identified in the output file by a value of '8' in the 'NUMBER' column or by a value of 's' in the 'LETTER' column. If the subject correctly responded to the target, this was identified by a value of '1' in the 'CORRECT=1' column. The number of accurate responses was calculated as the total number of records where 'CORRECT=1' had a value of '1'.
Time Frame: Baseline, 60 minutes and up to 120 minutes post treatment administration
Population: as for outcome 2
Measure: Median (Full Range); unit: Correct responses
Arm/Group | Paracetamol + Caffeine Combination (1000/130) | Paracetamol (1000) | Paracetamol + Caffeine Combination (500/65) | Paracetamol (500)
Number analyzed (Participants) | 45 | 45 | 75 | 75
Correct responses
  60 minutes | 10.0 [-9 to 34] | 6.0 [-35 to 66] | 8.0 [-9 to 45] | 5.5 [-27 to 82]
  120 minutes | 11.0 [-6 to 53] | 6.0 [-15 to 88] | 9.0 [-23 to 59] | 7.0 [-23 to 86]

9. Secondary Outcome: Change From Baseline in Mean Time of Accurate Responses to DAT Cognitive Test
Description: as for outcome 3
Time Frame: Baseline, 60 minutes and up to 120 minutes post treatment administration
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | Paracetamol + Caffeine Combination (1000/130) | Paracetamol (1000) | Paracetamol + Caffeine Combination (500/65) | Paracetamol (500)
Number analyzed (Participants) | 45 | 45 | 75 | 75
msec
  60 minutes | -3.0 (2.94) | 1.5 (2.94) | -4.4 (2.33) | -2.2 (2.28)
  120 minutes | -11.0 (3.00) | -5.3 (3.00) | -8.0 (2.37) | -4.6 (2.34)

10. Secondary Outcome: Change From Baseline in Number of Incorrect and Missed Responses to DAT Cognitive Test
Description: For the Divided Attention task, participants were required to respond on hearing the no. '8' in a continuous stream of numbers through headphones or seeing a letter 's' on screen. This was identified in the output file by a value of '8' in 'NUMBER' column or 's' in 'LETTER' column. If a subject responded incorrectly (pressed the response button at the wrong time), this was identified by a value of '-1' in 'CORRECT=1' column. The number of incorrect responses was calculated as the total no. of records where 'CORRECT=1' had a value of '-1'. If the subject missed a target (failed to press the response button on hearing the no. '8' or seeing the letter 's'), this was considered a missed response. The number of missed responses was calculated as the no. of records where there was a value of '8' in 'NUMBER' column or 's' in 'LETTER' column and a value of '0' in the 'CORRECT=1' column.
Time Frame: Baseline, 60 minutes and up to 120 minutes post treatment administration
Population: as for outcome 2
Measure: Mean (Standard Error); unit: incorrect and missed responses
Arm/Group | Paracetamol + Caffeine Combination (1000/130) | Paracetamol (1000) | Paracetamol + Caffeine Combination (500/65) | Paracetamol (500)
Number analyzed (Participants) | 45 | 45 | 75 | 75
incorrect and missed responses
  Incorrect responses at 60 minutes | -6.5 (1.02) | -4.2 (1.11) | -5.4 (0.87) | -3.3 (0.81)
  Incorrect responses at 120 minutes | -7.1 (1.01) | -4.9 (1.10) | -5.6 (0.86) | -5.0 (0.98)
  Missed responses at 60 minutes | -10.2 (1.27) | -7.6 (2.08) | -9.8 (1.19) | -6.2 (1.50)
  Missed responses at 120 minutes | -12.2 (1.54) | -9.1 (2.27) | -10.2 (1.43) | -7.8 (1.58)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of the treatment, and until 5 days following administration of the last dose of investigational product.
Arm/Group | Paracetamol + Caffeine Combination (1000/130) | Paracetamol (1000) | Paracetamol + Caffeine Combination (500/65) | Paracetamol (500)
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/45 | 0/74 | 0/75
Other Adverse Events (participants affected / at risk) | 0/46 | 0/45 | 0/74 | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.